CLINICAL TRIAL: NCT05361213
Title: Association Among Anthropometric Parameters and Neuromotor Behaviour in Neonates
Brief Title: Is There Any Correlation Among Neonates Anthropometry and Neuromotor Behaviour
Status: Completed | Type: Observational
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Professor, Maharishi Markandeshwar Institute of physiotherapy and rehabilitation, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Other Study IDs: MMDU/IEC/1924
Record Dates: First submitted 2022-03-31; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Cerebral Palsy, Autism or Other Neuromotor Behavior Abnormalities Correlation With Anthropometry
Keywords: Correlation; infants; muscles; weight; length
MeSH Terms: conditions — Cerebral Palsy; Autistic Disorder; Body Weight

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the association among anthropometric parameters and neuromotor behaviour in neonates for early identification and prediction of later neuromotor deficit.

DETAILED DESCRIPTION:
The association between anthropometric (birth weight, length and occipitofrontal circumference) measurement and hands-on measurement of above mentioned anthropometric dimensions and demographic dimension (bilateral forearm, midarm, calf and thigh) with neuromotor behaviour were explored.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born between ≥28 weeks and ≤ 42 weeks of gestation
* Birth weight between 1500 and 3000 grams
* Neonates are born under all the classifications of Fenton growth charts (SGA, AGA and LGA)
* Stable Hemodynamics
* Free from infection
* Stable vitals

Exclusion Criteria:

* Dermal conditions
* Chromosomal abnormalities
* History of surgery
* Neural tube defect
* Cardiac abnormally

Ages: 28 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Both term and preterm neonates from level III B NICU
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Neuromotor behaviour | at the baseline, single time on day first of assessment
  INFANIB scoring from 14- 70 score was documented
Demographic dimension | at the baseline demographic dimension measured, single time on day first
  Weight (kg) measured at baseline
Demographic dimensions | at the baseline demographic dimension measured, single time on day first
  length (cm) and occipitofrontal circumference (cm) measured at baseline
Anthropometric measurement | Anthropometry was documented single time on same day
  Both the sides forearm (cm), midarm (cm), thigh (cm) and calf circumference (cm) measurement

CONTACTS AND LOCATIONS:
Overall Officials: Asir John Samuel, PhD, Study Director — Maharshi Markandeshwar institute of physiotherapy and rehabilitation, mullana, ambala, india; Sunanda Bhowmik, MPT, Study Chair — Maharshi Markandeshwar institute of physiotherapy and rehabilitation, mullana, ambala, india; Jaishree Rai, (MPT), Principal Investigator — Maharshi Markandeshwar institute of physiotherapy and rehabilitation, mullana, ambala, india
Locations (1):
- Jaishree, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: Undecided